CLINICAL TRIAL: NCT04925804
Title: Unraveling Genetics of HypoPhosPhatasia (HPP Genetics) Observational Study
Brief Title: Unraveling Genetics of HypoPhosPhatasia (HPP Genetics)
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HPP genetics-2020
Record Dates: First submitted 2021-06-09; First posted 2021-06-14 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Hypophosphatasia
Keywords: Hypophosphatasia; HPP; non-ALPL
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on Dry Blood Spot (DBS) Filtercard (CentoCard®)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study to perform Whole Genome Sequencing in participants clinically suspected for HPP and negative for known pathogenic ALPL variants

DETAILED DESCRIPTION:
Hypophosphatasia (HPP) is a rare Inborn Error of Metabolism (IEM), characterized by low tissue-nonspecific isoenzyme of alkaline phosphatase (ALP) activity. Alkaline phosphatase (ALP) is crucial for osteoid mineralization. Its main substrate in bone is pyrophosphate (PPi), a natural inhibitor of mineralization. ALP cleaves pyrophosphate into its two phosphate moieties, which then become available to the mineralization process. This ALP deficiency results in accumulation of its substrates, mainly inorganic pyrophosphate (PPi), pyridoxal-5-phosphate (PLP), and phosphoethanolamine (PEA).

Beyond the bone and the Central Nervous System (CNS), ALP deficiency has an impact on a number of other organs and systems, resulting in a broad range of manifestations, including dental (premature tooth loss), muscular (muscle weakness, delayed walking, abnormal gait), rheumatic (calcium pyrophosphate deposition disease, fibromyalgia, fatigue, joint laxity), eye (calcifications), renal (nephrocalcinosis, kidney stones, renal failure), and gastrointestinal tract disturbance (gastroesophageal reflux).

The specific symptoms can vary greatly from one person to another, sometimes even among members of the same family. There are five major clinical forms of HPP (perinatal, infantile, childhood, adult, and odontohypophosphatasia), ranging from an extremely severe form that can cause stillbirth to a form associated with only premature loss of baby (deciduous) teeth, but no bone abnormalities.

The genetic reason of Hypophosphatasia is mainly caused by mutations in the ALPL gene, coding for the tissue nonspecific alkaline phosphatase isoenzyme. At least 397 distinct pathogenic variants (predominantly missense variants) were described to lead to low levels of the ALP enzyme. HPP can be inherited in an autosomal recessive (most perinatal and infantile forms) or autosomal dominant manner (typically the adult form and odontohypophosphatasia).

Since ALPL dependent prevalence is very low, while symptoms overlapping HPP are much more common, other primary - genetic - forms of HPP-like symptoms are to be sought and characterized.

The HPP genetics study aims to characterize the genetic background of HPP participants, who do not have pathogenic variant/s in the ALPL gene.

ELIGIBILITY:
* Informed consent is obtained from the participant or from the parent / legal guardian
* The participant is clinically suspected for HPP
* The participant does not have pathogenic variant/s in the ALPL gene
* The participant showed low alkaline phosphatase levels (age- and sex-adjusted) on at least two occasions at least a month apart based on the local laboratory reference range
* None of these conditions are present:

  * Celiac disease and
  * Clofibrate therapy and
  * Cleidocranial dysplasia and
  * Cushing's syndrome and
  * Hypothyroidism and
  * Massive Blood transfusion and
  * Milk-alkali syndrome and
  * Multiple myeloma and
  * Osteogenesis imperfecta, type II and
  * Pernicious or profound anemia and
  * Starvation and
  * Vitamin C deficiency and
  * Vitamin D intoxication and
  * Zinc deficiency and
  * Magnesium deficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The participant is clinically suspected for HPP with no pathogenic variant/s in the ALPL gene
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Genetic analysis (WGS) of participants clinically suspected for HPP | 6 months
  Analyis of Whole Genome Sequencing data in participants clinically suspected for HPP disease to characterize the genetic background of these 16 HPP subjects, who do not have pathogenic variant/s in the ALPL gene.

SECONDARY OUTCOMES:
Analysis and identification of genetic variants | 6 months
  Identification and validation of genetic variants in the selected cohort (16 WGS subjects; see Outcome 1) since ALPL dependent prevalence is very low, while symptoms overlapping HPP are much more common, other primary - genetic - forms of HPP-like symptoms are to be sought and characterized.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof. Dr., Study Chair — CENTOGENE GmbH
Locations (1):
- Universität Würzburg - Klinische Studieneinheit, Orthopädische Klinik, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
It is possible, but not determined, yet.

REFERENCES:
- [Derived] Seefried L, Petryk A, Del Angel G, Reder F, Bauer P. Whole genome sequencing in adults with clinical hallmarks of hypophosphatasia negative for ALPL variants. Mol Biol Rep. 2024 Sep 14;51(1):984. doi: 10.1007/s11033-024-09906-7. PMID 39276275